CLINICAL TRIAL: NCT03972904
Title: Effect of Light-Fat Rice® on Blood Glucose in Overweight/Obese Patients With Type 2 Diabetes Mellitus and Related Mechanisms
Brief Title: A Clinical Trial of Overweight/Obesity With Type 2 Diabetes
Acronym: ELFOOD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Hebei Dongfangyun Health Management Co.,Ltd (Unknown)
Responsible Party: Principal Investigator, Wei Chen, Peking Union Medical College Hospital,Clinical Nutrition Department,Chief Physician, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HS-1910
Record Dates: First submitted 2019-05-24; First posted 2019-06-04 (Actual); Last update posted 2020-09-28 (Actual); Status verified 2020-09

CONDITIONS: Diabetes Mellitus, Type 2; Overweight and Obesity
Keywords: Diabetes Mellitus,Type 2; Overweight; Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Overweight; Obesity

STUDY DESIGN:
Intervention Model Description: The diet will be administered by a professional physician (intervention group:Light-Fat Rice® combined with Active Peptide®; control group: staple food of equal energy containing a small amount of dietary fiber combined with comparable energy maltodextrin) with a lifestyle guidance,same in both groups, to assist in diabetes management. The method of taking the product can be divided into two parts.And a dynamic blood glucose transient monitor would be worn for all patients at the 3rd week to record the patients's dynamic blood glucose changes including preprandial, postprandial (every 15 minutes), before and after exercise (every 30 minutes).Besides these,the patients would be asked to record dietary and exercise diary for 3 days(including one weekend at least) each week also.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The Light-Fat Rice® group
  Interventions: Dietary Supplement: Light-Fat Rice® combined with Active Peptide®+ lifestyle guidance
- Control group (Placebo Comparator): The comparable energy staple food group
  Interventions: Dietary Supplement: A staple food of comparable energy containing a small amount of dietary fiber combined with a comparable energy maltodextrin + lifestyle guidance

INTERVENTIONS:
Dietary Supplement: Light-Fat Rice® combined with Active Peptide®+ lifestyle guidance — Subjects will be given the Light-Fat Rice® combined with Active Peptide® with a lifestyle guidance to assist diabetes management. The method of taking the product has two parts: 1.Light-Fat Rice®: 80g (1 pack) per day as a staple meal replacement, used as a separate staple food or mixed with other staple foods, taking 4 weeks; 2.Active Peptide®: 20g (2 packs) per day (1 pack each morning and evening), served with 300ml of 40°C warm water each time before meals and take it for 4 weeks.
  Arms: Intervention group
Dietary Supplement: A staple food of comparable energy containing a small amount of dietary fiber combined with a comparable energy maltodextrin + lifestyle guidance — A staple food of comparable energy containing a small amount of dietary fiber combined with a comparable energy maltodextrin (both produced by the same manufacturer) with a lifestyle guidance will be given by the professional to assist in diabetes management. The product is taken as follows: 1.equal-energy staple food containing a small amount of dietary fiber: 80g (1 pack) per day, used as an independent staple food or mixed with other staple foods, taking for 4 weeks; 2.equal-energy maltodextrin: 20g(2 packs) per day(1 pack each morning and evening),take it with 300ml of 40°C warm water for 4 weeks.
  Arms: Control group

SUMMARY:
In the previous intervention studies of Type 2 Diabetes Mellitus patients, changes in blood glucose and insulin resistance profiles before and after intervention indicated that different intervention methods had different effects on outcomes. Therefore, this study intends to explore the effect of the Light-Fat Rice®combined with Active Peptide® on the level of insulin resistance in overweight/obese diabetic patients and its effect on the outcome through a 4-week, randomized, double-blind, controlled clinical trial, further elucidating its intervention mechanism theoretically. The study predicts that dynamic blood glucose(mean blood glucose) and glycosylated albumin will significantly different between the control group and the intervention group.And insulin resistance levels, blood lipids and other indicators wil be improved, and the test group was superior to the control group.All of these will contribute to more scientific and effective Type 2 Diabetes Mellitus's management.

DETAILED DESCRIPTION:
The prevalence of Type 2 Diabetes Mellitus is increasing year by year in the world, causing harm to patients' health and making a huge consumption of medical expenses. Obesity is one of the most obvious risk factors for Type 2 Diabetes Mellitus. There are also many positive studies on nutritional intervention for the treatment of obese patients with Type 2 Diabetes Mellitus at home and abroad. The effect of nutritional meal replacement to relieve the disease has also been widely recognized.

Light-Fat Rice® is a new type of nutritious staple food taking rice, konjac, marine fish oligopeptide powder, inulin and yeast as raw material. Also,there is a protein solid beverage,Active Peptide®,containing soy protein isolate, soy peptide powder, oligofructose,water-soluble dietary fiber and other ingredients,such as multi-vitamin. When used together, it can provide balanced nutrition for the human body while satisfying low fat and high protein. In this study, a 4-week, randomized, double-blind, controlled clinical trial will be conducted to investigate the effects of Light-Fat Rice® combined with Active Peptide® intervention on insulin resistance in overweight/obese diabetic patients and their effects on prognosis,further explaining its intervention mechanism theoretically. Based on a previous review of similar literature studies, 60 of these patients will be enrolled and randomly assigned to the intervention and control groups at 1:1. Among them, the intervention group will be given 80g of Light-Fat Rice® staple food meal as an independent staple food or mixed in the staple food combined with 2 packs Active Peptide®, and the control group was given the same energy-equivalent staple food produced by the same manufacturer daily with 2 packs maltodextrin. Both groups are provided with a same lifestyle guidance by professional physicians based on the "Guidelines for the Prevention and Treatment of Type 2 Diabetes in China 2017", including reasonable diet, exercise guidance, and organization of health education.

ELIGIBILITY:
Inclusion Criteria:

1. Comply with the diagnostic criteria for type 2 diabetes in the 1999 WHO Diabetes Diagnosis and Classification Standard:

   Clear clinical record of fasting blood glucose (FPG) ≥ 7mmol / L or 75g OGTT（2h） ≥ 11.1mmol / L;
2. T2DM of duration > 1 year（diagnosis based on the 1999 WHO Diabetes Diagnosis and Classification Standard in China ）;
3. Body mass index: 25 kg/m2 < BMI ≤ 35kg/m2;
4. Men and women aged 18-75 years;
5. Volunteer to participate in the trial and sign the informed consent form .

Exclusion Criteria:

1. Acute cardiovascular and cerebrovascular events or myocardial infarction within previous 6 months;
2. Laboratory inspection:

   Liver function: AST and / or ALT ≥ 2.5 × ULN; Renal function: Cr>1.2×ULN;
3. People with severe gastrointestinal diseases, such as active peptic ulcer, intestinal obstruction, etc.;have a history of changes in the normal structure of the gastrointestinal tract;
4. Hypertensive patients with poor blood pressure control(blood pressure SBP≥160mmHg and / or DBP≥100mmHg);
5. Those with severe blood system diseases;
6. Combine other endocrine system diseases(such as hyperthyroidism or hypercortisolism);
7. Patients with stress or secondary blood glucose elevation(such as taking glucocorticoids);
8. Pregnant or lactating women,and women who are not willing to contraception during pregnancy or study;
9. Food or other drug abusers;
10. People who may be allergic to the test food;
11. Those who have participated in other food trials within 3 months;
12. Those who cannot co-operate with mental illness;
13. Other circumstances,which the researcher believes that it is not suitable for the group.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2019-06-20 (Actual); Primary Completion 2020-06-20 (Actual); Study Completion 2021-07-20 (Estimated)

PRIMARY OUTCOMES:
Dynamic blood glucose changes (average blood glucose) | week 3,week 4
  Patients will be exposed to a dynamic glycemic transient monitor from the 3rd week of the study period, worn for 2 weeks, and removed at the 4th week of follow-up. During the period of wearing, the patients will be required to record the dietary diary, preprandial and postprandial (every 15 minutes) blood glucose level (mmol/L) for 3-day period (including one day of the weekend)each week, and also select 3 days per week (including one day of the weekend) to record daily exercise, pre- and post-exercise (every 30 minutes) blood glucose levels (mmol/L) .
Insulin resistance index changes | Baseline time, week 4
  The patients will be subjected to two blood collections throughout the study, at baseline and at the 4th week of follow-up. The insulin resistance index is calculated as HOMA-IR=［plasma glucose（GLU,mmol/L）*serum insulin(mIU/L)］/22.5.

SECONDARY OUTCOMES:
Blood glucose control compliance rate | Baseline time, week 4
  The patients will be subjected to two blood collections throughout the study, at baseline and at the 4th week of follow-up. The glycemic control compliance rate will be compared using two fasting blood glucose values and expressed as a number (percentage).
Glycated albumin changes | Baseline time, week 4
  The patients will be subjected to two blood collections throughout the study, at baseline and at the 4th week of follow-up. The change in glycated albumin (GA%) will be compared with the values of two fasting blood samples, with a normal range of 10.8%-17.1%.

OTHER OUTCOMES:
Blood lipid changes | Baseline time, week 4
  The patients will be subjected to two blood collections throughout the study, at baseline and at the 4th week of follow-up. Changes in blood lipids (total cholesterol, mmol/L;triglycerides, mmol/L;high-density lipoprotein cholesterol, mmol/L; low-density lipoprotein cholesterol, mmol/L) will be compared using the values of two fasting blood samples. The normal range is 2.85-5.70 mmol/L for total cholesterol, 0.45-1.70 mmol/L for triglycerides, 1.42-11.29 mmol/L for high-density lipoprotein cholesterol, and 2.07-3.62 mmol/L for low-density lipoprotein cholesterol.
BMI changes | Baseline time, week 2,week 4
  Patients will be subjected to three body weight measurements throughout the study, baseline, week 2, and week 4 of follow-up,along with their height measurements at the start of the study. Both of the height and weight will be measured with a standard instrument and recorded in meters and kilograms respectively，following a requirement of accurating to two decimal places. And the weight and height will be combined to report in a form of BMI in kg/m^2.The changes in BMI before and after the study will be expressed as mean ± SD.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Chen, M.D., Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Dongcheng district，Peking union medical college hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
The following data will be shared at the end of the study: demographic data, current medical history, past history; physical examination data collected at 3 visits, including heart rate, blood pressure, height, weight, waist circumference, hip circumference, grip strength, and human body Ingredients, etc.; previous physical examination data provided at baseline such as abdominal ultrasound; laboratory tests such as insulin levels, blood lipid levels, urinary protein levels collected at baseline and 4th week of follow-up; dietary and exercise diaries as well as the dynamic blood sugar changes along with these, etc.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: The data is expected to be available after June，20, 2020 and can be used forever.
Access Criteria: The information should be used for academic research, medical communication, etc., and is prohibited from being used for commercial gain.

REFERENCES:
- [Background] Ryan DH, Espeland MA, Foster GD, Haffner SM, Hubbard VS, Johnson KC, Kahn SE, Knowler WC, Yanovski SZ; Look AHEAD Research Group. Look AHEAD (Action for Health in Diabetes): design and methods for a clinical trial of weight loss for the prevention of cardiovascular disease in type 2 diabetes. Control Clin Trials. 2003 Oct;24(5):610-28. doi: 10.1016/s0197-2456(03)00064-3. PMID 14500058
- [Background] Leslie WS, Ford I, Sattar N, Hollingsworth KG, Adamson A, Sniehotta FF, McCombie L, Brosnahan N, Ross H, Mathers JC, Peters C, Thom G, Barnes A, Kean S, McIlvenna Y, Rodrigues A, Rehackova L, Zhyzhneuskaya S, Taylor R, Lean ME. The Diabetes Remission Clinical Trial (DiRECT): protocol for a cluster randomised trial. BMC Fam Pract. 2016 Feb 16;17:20. doi: 10.1186/s12875-016-0406-2. PMID 26879684
- [Background] Lean ME, Leslie WS, Barnes AC, Brosnahan N, Thom G, McCombie L, Peters C, Zhyzhneuskaya S, Al-Mrabeh A, Hollingsworth KG, Rodrigues AM, Rehackova L, Adamson AJ, Sniehotta FF, Mathers JC, Ross HM, McIlvenna Y, Stefanetti R, Trenell M, Welsh P, Kean S, Ford I, McConnachie A, Sattar N, Taylor R. Primary care-led weight management for remission of type 2 diabetes (DiRECT): an open-label, cluster-randomised trial. Lancet. 2018 Feb 10;391(10120):541-551. doi: 10.1016/S0140-6736(17)33102-1. Epub 2017 Dec 5. PMID 29221645
- [Background] Lean MEJ, Leslie WS, Barnes AC, Brosnahan N, Thom G, McCombie L, Peters C, Zhyzhneuskaya S, Al-Mrabeh A, Hollingsworth KG, Rodrigues AM, Rehackova L, Adamson AJ, Sniehotta FF, Mathers JC, Ross HM, McIlvenna Y, Welsh P, Kean S, Ford I, McConnachie A, Messow CM, Sattar N, Taylor R. Durability of a primary care-led weight-management intervention for remission of type 2 diabetes: 2-year results of the DiRECT open-label, cluster-randomised trial. Lancet Diabetes Endocrinol. 2019 May;7(5):344-355. doi: 10.1016/S2213-8587(19)30068-3. Epub 2019 Mar 6. PMID 30852132
- [Background] Laws R; Counterweight Project Team. A new evidence-based model for weight management in primary care: the Counterweight Programme. J Hum Nutr Diet. 2004 Jun;17(3):191-208. doi: 10.1111/j.1365-277X.2004.00517.x. PMID 15139891